CLINICAL TRIAL: NCT05501938
Title: Randomized Controlled Trial: Physical Exam Indicated Cerclage in Singleton Gestation 24 Weeks to 25 Weeks and 6 Days Gestation
Brief Title: Physical Exam Indicated Cerclage in Singleton Gestation 24 Weeks to 25 Weeks and 6 Days Gestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Craig Zelig, Director of Maternal Fetal Medicine; MFM Fellowship Director, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6456
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Intervention (cerclage) and control (no-cerclage) to reduce/prevent preterm delivery in those with a dilated cervix between 24w0d and 25w6d
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerclage (Experimental): Perform physical exam indicated cerclage between 24w0d to 25w6d
  Interventions: Procedure: Physical Exam Indicated Cerclage
- Control (No Intervention): No intervention; routine monitoring in pregnancy for preterm delivery

INTERVENTIONS:
Procedure: Physical Exam Indicated Cerclage — Transvaginal cervical cerclage
  Arms: Cerclage

SUMMARY:
RCT assessing preterm delivery rate in singleton pregnancies having a physical-exam indicated cerclage placed between 24 weeks and 25 weeks and 6 days. Patients randomized to either cerclage intervention or routine standard of care (no cerclage).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women 18 years of age or older
2. Nulliparous patient, has not had a preterm to term delivery
3. Singleton pregnancy
4. English or Spanish speaking
5. Asymptomatic cervical dilation between 1- 2 cm, without visible membranes beyond the external cervical os and without any evidence of infection, active labor or active bleeding between 24 0/7 and 25 6/7 weeks gestation

Exclusion Criteria:

1. Twin or higher order multi-fetal gestation
2. Multiparous patient, has had one or more preterm to term deliveries
3. Cervical dilation more than 2 cm either at the beginning of the study or any time during the study
4. Amniotic membranes prolapsed beyond the external os
5. Fetal reduction procedure performed during current pregnancy
6. Ruptured membranes prior to randomization
7. Major fetal structural anomaly
8. Fetal chromosomal abnormality, suspected or confirmed with additional genetic testing
9. Cerclage already in place for other indication
10. Active vaginal bleeding
11. Suspicion of chorioamnionitis
12. Placenta previa
13. Painful regular uterine contractions
14. History of preterm birth before 37 weeks gestation
15. Non-English or non-Spanish speaking

    a. Given that the study is explained in person and consent forms are written in English, there is no guarantee that the study will be explained correctly when using a phone translator. The same is true if the current English consent form were to be translated into a language other than English. There is no way to confirm that the integrity of the study is being upheld by using translating services. If the integrity of the study is not upheld, then this poses harm to the patient.
16. Women under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-08-11 (Estimated); Primary Completion 2023-08-11 (Estimated); Study Completion 2023-08-11 (Estimated)

PRIMARY OUTCOMES:
Preterm Delivery Rate | 1 Year
  Compare preterm delivery rate between women receiving cerclage intervention between 24w0d and 25w6d vs those not receiving cerclage during this gestational age period

SECONDARY OUTCOMES:
Neonatal Outcomes | 1 Year
  Rate of neonatal outcomes compared between the two groups ( NICU length of stay, neonatal death, neonatal disease (bronchopulmonary dysplasia, Necrotizing enterocolitis, Intraventricular hemorrhage, Respiratory distress syndrome, Retinopathy of prematurity, sepsis, death)

OTHER OUTCOMES:
Cerclage Surgical Complications | 1 year
  Rate of cerclage complications (intra-operative PPROM, hemorrhage, need for blood transfusion, cervical or vaginal laceration

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided